CLINICAL TRIAL: NCT06263140
Title: A Study of Vitamin D Levels in Patients With Non-immediate Drug Hypersensitivity, Case-control Study
Brief Title: Vitamin D Levels in Non-immediate Drug Hypersensitivity Case-control Study
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Other Study IDs: Chula-ARC 001/21
Record Dates: First submitted 2022-02-09; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2022-02

CONDITIONS: Stevens-Johnson Syndrome; Drug Reaction With Eosinophilia and Systemic Symptom; Maculopapular Exanthem; Vitamin D Deficiency; Drug-Induced Rash
Keywords: vitamin D; Stevens-Johnson Syndrome; Drug Reaction with Eosinophilia and Systemic Symptom; Maculopapular Exanthem; Drug Allergy; Drug Hypersensitivity
MeSH Terms: conditions — Stevens-Johnson Syndrome; Drug Hypersensitivity Syndrome; Drug Eruptions; Vitamin D Deficiency; Drug Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1. Patients diagnosed with drug-induced severe non-immediate cutaneous reactions: Stevens-Johnson syndrome (SJS)/toxic epidermal necrolysis (TEN), drug reaction with eosinophilia and systemic symptom (DRESS), acute generalized exanthematous pustulosis (AGEP)
- 2. Patients diagnosed with drug-induced non-severe non-immediate cutaneous reactions: Maculopapular exanthem (MPE), fixed drug eruption (FDE)
- 3. Subjects who tolerated drugs potentially causing severe non-immediate cutaneous reactions: Studied drug groups matched patients in group 1
- 4. Subjects who tolerated drugs potentially causing non-severe non-immediate cutaneous reactions: Studied drug groups matched patients in group 2

SUMMARY:
Serum vitamin D levels in drug-induced non-immediate reactions

DETAILED DESCRIPTION:
The study of serum vitamin D levels in patients presented with drug-induced non-immediate cutaneous adverse reactions compared to those in drug-tolerant control subjects

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with SJS/TEN, DRESS, AGEP, MPE, or FDE as mentioned above

Exclusion Criteria:

* Reactions from drugs with known strong genetic predispositions (allopurinol, carbamazepine, abacavir)
* Receiving vitamin D supplement

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases: Subjects who develop drug-induced non-immediate cutaneous reactions
  Controls: subjects who can tolerate similar drug groups without allergic reactions
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Serum vitamin D levels | At baseline
  Serum vitamin D levels at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jettanong klaewsongkram, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand